CLINICAL TRIAL: NCT06345014
Title: A Multicenter, Randomized, Placebo-controlled, Double-blind, Phase 4 Study to Evaluate the Efficacy and Safety of OM-89 in Patients With Recurrent Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS)
Brief Title: The Efficacy and Safety of OM-89 in Patients With Recurrent Chronic Prostatitis/Chronic Pelvic Pain Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AJU Pharm Co., Ltd. (Industry)
Collaborators: OM Pharma SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23CP40803
Record Dates: First submitted 2024-03-24; First posted 2024-04-03 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome; Chronic Prostatitis; Chronic Pelvic Pain Syndrome
Keywords: CP/CPPS; Chronic Prostatitis; Chronic Pelvic Pain Syndrome
MeSH Terms: conditions — Prostatitis | interventions — OM 89

STUDY DESIGN:
Intervention Model Description: Once a subject voluntarily gives written consent to participate in this study, a screening test will be conducted to evaluate their eligibility. Subjects determined to be eligible to participate in the study on Visit 2 (baseline) will be enrolled, randomized 1:1 either to the test group (OM-89 [Uro-Vaxom® Capsule]) or the control group (placebo of OM-89) and administered the investigational product for 26 weeks.
  In parallel, an alpha blocker (alfuzosin 10 mg) will be administered for the first 13 weeks as a background treatment, followed by the placebo of alfuzosin until Week 26. The efficacy and safety will be checked until Week 52 from the start of the treatment for all subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Background treatment - Xatral® XL Tab. 10 mg (alfuzosin hydrochloride): With the treatment of the investigational product, it will be administered for the first 13 weeks (Administration of the placebo will be continued to maintain the treatment compliance and blinding for the rest 13 weeks).
  After week 13, Background treatment will be blinded for subject only until end of treatment period(Week 26).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Drug: OM-89 (Uro-Vaxom® Capsule 60 mg (6 mg as a freeze-dried bacterial lysate)) (Experimental): - OM-89 (Uro-Vaxom® Capsule 60 mg (6 mg as a freeze-dried bacterial lysate)) Oral administration of the investigational product (OM-89 [Uro-Vaxom® Capsule] or the placebo) once a day.
  Interventions: Drug: OM-89 [Uro-Vaxom® Capsule]
- Comparator: (Placebo Comparator): - Placebo of Uro-Vaxom® Capsule Oral administration of the investigational product (OM-89 [Uro-Vaxom® Capsule] or the placebo) once a day.
  Interventions: Drug: OM-89 Placebo [Uro-Vaxom® Capsule Placebo]

INTERVENTIONS:
Drug: OM-89 [Uro-Vaxom® Capsule] — Oral administration of the investigational product (OM-89 [Uro-Vaxom® Capsule] or the placebo) once a day
  Other Names: Test Group(OM-89 group)
  Arms: Study Drug: OM-89 (Uro-Vaxom® Capsule 60 mg (6 mg as a freeze-dried bacterial lysate))
Drug: OM-89 Placebo [Uro-Vaxom® Capsule Placebo] — Oral administration of the investigational product(Placebo of Uro-Vaxom® Capsule)
  Other Names: Placebo Group(OM-89 Placebo group)
  Arms: Comparator:

SUMMARY:
This study is planned to Evaluate the Efficacy and Safety of OM-89 in Patients with Recurrent Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS)

DETAILED DESCRIPTION:
This clinical study is designed as a multicenter, randomized, placebo-controlled, double-blind, phase 4 study to evaluate the efficacy and safety of the combination therapy of Uro-Vaxom® Capsule and alfuzosin in patients with recurrent chronic prostatitis.

Once a subject voluntarily gives written consent to participate in this study, a screening test will be conducted to evaluate their eligibility. Subjects determined to be eligible to participate in the study on Visit 2 (baseline) will be enrolled, randomized 1:1 either to the test group (OM-89 [Uro-Vaxom® Capsule]) or the control group (placebo of OM-89) and administered the investigational product for 26 weeks.

In parallel, an alpha blocker (alfuzosin 10 mg) will be administered for the first 13 weeks as a background treatment, followed by the placebo of alfuzosin until Week 26.

The efficacy and safety will be checked until Week 52 from the start of the treatment for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male adults aged ≥19 to ≤55 at the time of obtaining the written consent
* Those who have t pain or discomfort in the pelvic or genital area
* NIH-CPSI (the National Institutes of Health Chronic Prostatitis Symptom Index) ≥ 15 in total score
* voluntarily signed the informed consent form to participate in this study

Exclusion Criteria:

* Prostate specific antigen (PSA) ≥ 4.0 ng/ml at Visit 1 (screening)
* Received a prostate biopsy, surgery, or treatment within 12 weeks before Visit 1 (screening)
* Past or current medical history as Herpes infection treatment within 1 year before the Screening,Treatment for genital infections or sexually transmitted diseases and History of urogenital tumors.
* Those who have a medication history of the drugs(Drugs or health functional food, Health functional foods that affect prostate function etc)or have a plan to receive them during the study at Visit 1

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 332 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
NIH-CPSI total score | WEEK 4, 13, 26, 39, 52
  National Institute of Health Chronic Prostatitis Symptom Index (Minimum Score = 0 to Maximum Score=43, Higher score means worse outcome)

SECONDARY OUTCOMES:
NIH-CPSI domain score | WEEK 4, 13, 26, 39, 52
  pain, urinary symptoms, and effect on quality of life (Higher score means worse outcome)
Subject and Investigator's Global Assessment | WEEK 4, 13, 26, 39, 52
  Subject and Investigator's Global Assessment (Higher score means worse outcome, Very dissatisfied=1 to very satisfied=5)

CONTACTS AND LOCATIONS:
Locations (1):
- AJU Pharm Co., Ltd., Seoul, South Korea